CLINICAL TRIAL: NCT06319183
Title: The Regulatory Function of Inhaled Asthma Medication Salbutamol on Thermogenesis
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Tongji University (Other)
Responsible Party: Principal Investigator, Junkun Jiang, postdoctor, Tongji University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023tjdxsy045
Record Dates: First submitted 2024-03-13; First posted 2024-03-19 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Effect of Asthma Medication Salbutamol on Obesity
MeSH Terms: interventions — Albuterol

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Salbutamol (Experimental)
  Interventions: Drug: Salbutamol

INTERVENTIONS:
Drug: Salbutamol — We will recruit at least 15 male and 15 female volunteers, dividing study participants into two groups based on sex. Before administration, the temperature of the brown adipose tissue area in the scapular region of participants will be recorded using an infrared thermometer. Subsequently, participants will inhale the asthma medication salbutamol according to the safe dosage requirements (100ug). Eight hours later, the temperature changes in the brown adipose tissue area in the scapular region will be detected using an infrared thermometer. During the 8-hour waiting period, the participants' heart rate and blood pressure will be monitored; finally, we will draw 1 milliliter of venous blood from the arm of the participants for blood component analysis. The single trial process will last up to 8 hours, with no follow-up required.

SUMMARY:
In recent years, obesity and its complications have severely threatened human health. Given the limited options for obesity treatment currently available, there is an urgent need to develop new drugs and therapeutic methods to alleviate patient suffering.

Mammalian adipose tissue is primarily divided into energy-storing white fat and energy-consuming brown fat. Physical activity, exposure to cold, and other factors induce the transformation of white fat into energy-consuming brown fat, a process known as adipose tissue browning. The occurrence of adipose tissue browning increases the body's energy expenditure and dissipates it in the form of heat, effectively mitigating the onset of obesity. Therefore, the regulatory mechanism of adipose tissue browning has become an important potential target for obesity treatment.

The main component of asthma medication is the β2 adrenergic receptor agonist, which can act on GPCR receptors on the surface of the tracheal smooth muscle through inhalation, causing bronchial dilation and thereby alleviating asthma symptoms. Preliminary experimental results have shown that pulmonary epithelial cells can secrete protein factors that regulate the browning process of adipose tissue, and the expression of these secretory factors is regulated by the cell surface GPCR receptor signaling pathway. Therefore, our goal is to validate the regulatory effect of the asthma medication salbutamol on adipose tissue browning through inhalation administration in humans, establishing a new function for asthma medication in obesity treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 20-40 years, with at least 15 males and 15 females;
2. After administering the drug, the heart rate, blood pressure, and blood components of the subjects will be tested;
3. No history of asthma or diagnosed with bronchial asthma according to the "Chinese Guidelines for the Prevention and Treatment of Bronchial Asthma (2016 Edition)," and currently still in the persistent phase;
4. During the lead-in period and treatment period of the study, able to discontinue the study drug and other beta-receptor agonist medications used for treating asthma (such as inhaled long-acting beta-receptor agonists);
5. Subjects who agree to participate in this clinical trial and sign a written informed consent form.

Exclusion Criteria:

1. Subjects with clinically significant major pulmonary diseases;
2. Subjects with other diseases associated with elevated eosinophil counts;
3. Individuals allergic to Salbutamol;
4. Individuals allergic to fluorocarbons used as propellants;
5. Patients with cardiovascular dysfunction, insufficient coronary artery supply, hypertension, diabetes, and hyperthyroidism;
6. Individuals allergic to other adrenergic receptor agonists;
7. Women who are pregnant, breastfeeding, or planning to become pregnant in the near future;
8. Individuals with rare hereditary digestive system diseases - lactose intolerance, lactase deficiency, or glucose-galactose malabsorption;
9. Other reasons deemed by the researcher as inappropriate for participation in the trial.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-03 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Temperature of Scapular Region | Eight hours
  The temperature of the brown adipose tissue area in the scapular region of participants will be recorded before and after salbutamol administration using an infrared thermometer

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: After the related articles are published, these data will be made available to other researchers for reference.